CLINICAL TRIAL: NCT06403579
Title: THE EFFECT OF VIRTUAL REALITY APPLICATION ON PAIN, ANXIETY, AND COMFORT DURING CURETTAGE/DILATATION: A RANDOMIZED CONTROLLED TRIAL
Brief Title: THE EFFECT OF VIRTUAL REALITY APPLICATION ON PAIN, ANXIETY, AND COMFORT DURING CURETTAGE/DILATATION
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, seda karaçay yıkar, Assistant professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 142-16
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Bleeding;Post D&C; PAIN, ANXIETY, AND COMFORT
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality application (Experimental): Experimental: virtual reality application virtual reality goggles will be implemented.
  Interventions: Device: virtula reality goggles
- control (Sham Comparator): No Intervention: control group no intervention will be made
  Interventions: Device: virtula reality goggles

INTERVENTIONS:
Device: virtula reality goggles — no intervention
  Other Names: control

SUMMARY:
The problems experienced by women at the stage of deciding to have a miscarriage, during and after miscarriage differ and their anxiety levels vary. It was determined that women experienced fear, thinking that they would sin, guilt, regret and indecision at the stage of deciding to abort. methods are used to relieve the pain and anxiety caused by interventional procedures in patients in direct proportion to the development of technology. Virtual reality (VR), one of these methods, is an innovative, up-to-date and unique application, combining reality and imagination with fictional technology.There is no study in the literature on the application of SG during curettage/dilatation procedure. This study was conducted to determine the effect of SG application on pain anxiety and comfort during curettage/dilatation procedure.

ELIGIBILITY:
Inclusion Criteria:

* 15-49 years old,
* Termination ordered,
* Can speak and understand Turkish,

Exclusion Criteria:

* - Cognitive, effective and without any problem preventing communication,
* No psychiatric problems,
* Diagnosed with epilepsy (due to the risk that SG glasses may trigger epileptic seizures),
* Women who volunteer to participate in the study will be recruited.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women will be included
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
virtual reality application | at 1 hour after curettage
  virtual reality application reduces women's pain scores 0-5 points
virtual reality application | at 1 hour after curettage
  virtual reality application reduces women's anxiety scores 20-39 points
virtual reality application virtual reality application | at 1 hour after curettage
  virtual reality application reduces women's anxiety scores 24-144 points

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Karaçay Yıkar, Adana, Sarıcam, Turkey (Türkiye)